CLINICAL TRIAL: NCT02458235
Title: A Phase II Study of Risk-adapted Donor Lymphocyte Infusion and Azacitidine for the Prevention of Hematologic Malignancy Relapse Following Allogeneic Stem Cell Transplantation
Brief Title: Donor Lymphocyte Infusion With Azacitidine to Prevent Hematologic Malignancy Relapse After Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Hellman Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140813; NCI-2015-02240 (Registry Identifier: University of California, San Francisco)
Record Dates: First submitted 2015-01-05; First posted 2015-06-01 (Estimated); Results first posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Acute Myelogenous Leukemia; Acute Lymphoid Leukemia; Juvenile Myelomonocytic Leukemia; Myelodysplastic Syndrome
Keywords: pediatric leukemia myelodysplastic syndrome azacitidine
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelomonocytic, Juvenile; Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Azacitidine/donor lymphocyte infusion (Experimental): Patients will be stratified according to risk categories (low, standard and high), defined by GVHD status, mixed versus full donor chimerism, and positive versus negative Minimal Residual Disease (MRD) results. Patients will receive up to 7 cycles of low-dose azacitidine (40mg/m2 IV/SC daily x 4 days) at 6 weekly intervals, except for low risk ALL patients who may not receive treatment after withdrawal of immunosuppression. Standard risk patients will receive an additional 6 cycles of azacitidine alone. High risk patients will receive an additional 6 cycles of azacitidine plus escalating DLI.
  Interventions: Drug: azacitidine; Biological: donor lymphocyte infusion

INTERVENTIONS:
Drug: azacitidine — 40mg/m2 IV/SC daily x 4 days, maximum of 7 cycles at 6 weekly intervals
  Other Names: Vidaza®, Ladakamycin
Biological: donor lymphocyte infusion — For patients with cells available for DLI who are in the high risk group and do not have graft-versus-host disease (GVHD), DLI will be adminstered on day 5 of each cycle.

SUMMARY:
The goal of this study is to determine whether post-transplant consolidation with azacitidine combined with donor lymphocyte infusion (DLI) is a safe and effective approach for the prevention of relapse in pediatric and young adult patients with hematologic malignancies who have undergone hematopoietic stem cell transplantation (HSCT).

DETAILED DESCRIPTION:
This is a phase II single-arm trial of azacitidine (IV or SC) in combination with escalating donor lymphocyte infusion (DLI). Patients will be enrolled on the study by day +28 +/- 7 post-transplant, prior to withdrawal of immunosuppression or administration of donor lymphocyte infusion (DLI). They will have donor chimerism and minimal residual disease (MRD) testing from peripheral blood (PB) and bone marrow (BM) on day +28 ± 7. Patients will be stratified according to risk categories (low, standard and high), defined by GVHD status, mixed versus full donor chimerism, and positive versus negative MRD results. Depending on risk assessment, immunosuppression will be tapered according to standard or fast schedules, and patients (with the exception of low-risk ALL patients) will receive one cycle of low-dose azacitidine (40mg/m2 IV/SC daily x 4 days). After tapering immunosuppression, chimerism will be repeated and patients will receive up to 6 additional cycles of low-dose azacitidine, depending on risk assessment. For patients who meet criteria for high risk of relapse, azacitidine will be combined with escalating doses of DLI for a maximum of 7 cycles in total. Risk and safety assessments, including routine laboratory parameters, donor chimerism, minimal residual disease, and GHVD activity will be assessed following each cycle. Chimerism and minimal residual disease testing will be repeated every cycle by peripheral blood (PB), and bone marrow (BM) will be tested every other cycle. Patients will be followed by laboratory monitoring and physician evaluation prior to each cycle, and will be followed for two years post-transplant to study toxicity and GVHD outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 0 - 29.9 years undergoing allogeneic peripheral blood stem cell transplant
* Patients with acute myelogenous leukemia (AML) or acute lymphoblastic leukemia (ALL)
* Patients with juvenile myelomonocytic leukemia (JMML)
* Patients with myelodysplastic syndrome (MDS)

Exclusion Criteria:

* Patients who have had a prior transplant.
* Patients with Fanconi anemia or other cancer-predisposition syndromes
* Patients with expected survival <12 weeks
* Lansky score <60%

Max Age: 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2015-06-02 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C Dvorak, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Justin T. Wahlstrom, Biljana N. Horn, Carol Fraser-Browne, Rebecca Hoeweler, Ying Lu, Alexis Melton, Jennifer Willert, Christopher C. Dvorak; Azacitidine Administration Following Hematopoietic Stem Cell Transplantation Is Safe and Feasible in Children with Acute Leukemia. Blood 2016; 128 (22): 4805. https://doi.org/10.1182/blood.V128.22.4805.4805

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Azacitidine/Donor Lymphocyte Infusion
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Azacitidine/Donor Lymphocyte Infusion
Number analyzed (Participants) | 17
Age, Customized [Count of Participants; unit: Participants]
  0-9 years | 7
  10-19 years | 9
  20-29 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Relapse Rate
Description: Relapse rate will be estimated using a percentage of participants who relapsed. It is assumed that the rate of relapse in pediatric acute leukemia post-transplant would be 40%, azacitidine +/- Donor Lymphocyte Infusion (DLI) would reduce the 2-year relapse rate by approximately 40% to a rate of 25%.
Time Frame: Up to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Azacitidine/Donor Lymphocyte Infusion
Number analyzed (Participants) | 17
percentage of participants | 23.5

2. Primary Outcome: Frequency of System Specific Grade 3 or Higher Treatment-related Adverse Events
Description: Frequency of system specific adverse events of interest include renal, hepatic, cardiac, pulmonary, or neurologic toxicities. Toxicities will be graded using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Azacitidine/Donor Lymphocyte Infusion
Number analyzed (Participants) | 17
Participants | 0

3. Primary Outcome: Proportion of Participants With Acute and Chronic Graft Versus Host Disease (GVHD)
Description: Proportion of participants with Grade 3-4 acute GVHD and moderate to severe chronic GVHD will be reported.
Time Frame: Up to 2 years
Measure: Number; unit: proportion of participants
Arm/Group | Azacitidine/Donor Lymphocyte Infusion
Number analyzed (Participants) | 17
proportion of participants
  Acute GVHD | 0.176
  Moderate to severe chronic GVHD | 0.411

4. Primary Outcome: Proportion of Participants With Serious Infection
Description: The proportion of participants will be reported for Grade 3-4 invasive fungal infection or disease caused by viral infections
Time Frame: Up to 2 years
Measure: Number; unit: proportion of participants
Arm/Group | Azacitidine/Donor Lymphocyte Infusion
Number analyzed (Participants) | 17
proportion of participants | 0.41

5. Primary Outcome: Proportion of Participants With Severe Hematologic Toxicity Including Graft Failure
Description: The proportion of participants will be reported for Grade 4 severe hematologic toxicities including graft failure
Time Frame: Up to 2 years
Population: No participants experienced a severe hematologic toxicity including graft failure
Measure: Number; unit: proportion of participants
Arm/Group | Azacitidine/Donor Lymphocyte Infusion
Number analyzed (Participants) | 17
proportion of participants | 0.00

6. Primary Outcome: Number of Participants Whom Had >2 Dose Reductions for Any Reason
Description: The number of participants whom had greater than 2 dose reductions for any reason.
Time Frame: Up to 2 years
Measure: Number; unit: participants
Arm/Group | Azacitidine/Donor Lymphocyte Infusion
Number analyzed (Participants) | 17
participants | 0

7. Secondary Outcome: Median Relapse-free Survival
Description: Release-free survival rate is defined as the median length of time after beginning treatment that the participant survives without progression or relapse, reported in months
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Azacitidine/Donor Lymphocyte Infusion
Number analyzed (Participants) | 17
months | 22 [1 to 24]

8. Secondary Outcome: Median Time to Relapse
Description: Time to relapse is defined as the length of time after beginning treatment until the participant has experienced a relapse in disease, measured in months.
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Azacitidine/Donor Lymphocyte Infusion
Number analyzed (Participants) | 17
months | 3 [1 to 17]

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Azacitidine/Donor Lymphocyte Infusion
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 10/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azacitidine/Donor Lymphocyte Infusion (N=17)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Immune system disorders - Other (Immune system disorders) | 3 (3)
Fever (General disorders) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Cardiac disorders - Other (Cardiac disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 (1)
Elevated transaminases (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azacitidine/Donor Lymphocyte Infusion (N=17)
Acute GVHD (Investigations) | 3 (3)
Adrenal insufficiency (Endocrine disorders) | 3 (3)
Anisocoria (Eye disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Cholestatic liver disease (Hepatobiliary disorders) | 1 (1)
Chronic GVHD (Investigations) | 7 (7)
Chronic Pain (General disorders) | 3 (3)
Conductive Hearing Loss (Ear and labyrinth disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Cytomegalovirus (CMV) viremia (Infections and infestations) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Electrolyte Abnormality (Investigations) | 1 (1)
Emotional disturbance (Psychiatric disorders) | 1 (1)
Epileptic seizures (Nervous system disorders) | 1 (1)
Fever (General disorders) | 4 (4)
Foreskin adhesions (Reproductive system and breast disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Headaches (Nervous system disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Human Herpesvirus 6 (HHV-6) viremia (Infections and infestations) | 1 (1)
Human Metapneumovirus (hMPV) (Infections and infestations) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Iron overload (Metabolism and nutrition disorders) | 4 (4)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Neuropathy (Vascular disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2)
Post Transplant Immunodeficiency (Investigations) | 17 (17)
Pseudoseizures (Nervous system disorders) | 1 (1)
Pulmonary aspergillosis (Infections and infestations) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Weight Loss (Investigations) | 2 (2)
Abnormal alanine aminotransferase (ALT) and aspartate aminotransferase (AST) (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2015-05-05): https://cdn.clinicaltrials.gov/large-docs/35/NCT02458235/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-11-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT02458235/Prot_SAP_001.pdf